CLINICAL TRIAL: NCT04010695
Title: Validation of Diagnostics to Identify Glucose-6-phosphate Dehydrogenase Activity in the US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: G6PD Validation Seattle
Record Dates: First submitted 2019-05-21; First posted 2019-07-08 (Actual); Results first posted 2021-08-26 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2021-06

CONDITIONS: G6PD Deficiency
Keywords: G6PD deficiency
MeSH Terms: conditions — Glucosephosphate Dehydrogenase Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- G6PD Diagnostic Testing (Other): Participants provided whole blood samples as well as fingerstick capillary blood samples.
  At the clinic site lab, study staff conducted the SD Biosensor point-of-care G6PD test and the point-of-care HemoCue Hb test on both finger stick blood and whole blood samples.
  At the reference laboratory, G6PD activity was measured from whole blood samples using the Pointe Scientific G6PD reference assay and hemoglobin was measured using a hematology analyzer.
  Interventions: Diagnostic Test: SD Biosensor G6PD Analyzer; Diagnostic Test: Pointe Scientific Test Kit; Diagnostic Test: HemoCue System

INTERVENTIONS:
Diagnostic Test: SD Biosensor G6PD Analyzer — The SD Biosensor G6PD Analyzer is designed to measure the quantitative determination of total hemoglobin concentration and G6PD enzymatic activity in fresh human whole blood specimens based on reflectometry assays in a point-of-care setting. The test is intended to aid in the identification of people with G6PD deficiency. The test is currently not licensed for use in the US and is considered an investigational product.
Diagnostic Test: Pointe Scientific Test Kit — The Pointe Scientific test kit will serve as the reference assay to assess G6PD activity. Its intended use is for the quantitative, kinetic determination of G6PD in blood at 340 nm.
Diagnostic Test: HemoCue System — The HemoCue hemoglobin (Hb) 201+ system is designed for quantitative point-of-care whole blood hemoglobin determination in primary care using a specially designed analyzer, the HemoCue Hb 201+ Analyzer, and specially designed microcuvettes, the HemoCue Hb 201+Microcuvettes.

SUMMARY:
The primary objective of this study is to assess the accuracy of the SD Biosensor STANDARD G6PD Analyzer in measuring G6PD activity when used by trained health care workers.

DETAILED DESCRIPTION:
This is a cross-sectional diagnostic accuracy study with up to 250 participants with a goal of obtaining 20 deficient and 20 intermediate samples. The clinic will recruit and consent study participants. Clinic staff will draw 3 whole blood samples and obtain finger stick capillary blood.

G6PD activity is reported in terms of grams of hemoglobin (Hb), hence the hemoglobin concentration must be measured.

Clinic staff will perform the investigational Standard Diagnostics (SD) Biosensor point-of-care (POC) test for glucose-6-phosphate dehydrogenase (G6PD) deficiency and a HemoCue® hemoglobin test on finger stick capillary blood and on the venous blood samples.

Another venous blood sample will be sent to a clinical laboratory improvement amendments (CLIA)-certified laboratory for reference testing by the gold standard assays:

* G6PD measurement by spectrophotometry using the Pointe Scientific G6PD reference assay
* hemoglobin measurement by a hematology analyzer

Individuals identified as G6PD deficient with the reference test will be notified of their results by the clinic and referred to their physician for follow-up.

ELIGIBILITY:
Inclusion Criteria:

-Willingness to provide consent

Exclusion Criteria:

-Blood transfusion in the past 90 days by self-report

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Kublin, MD, MPH, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchison Prevention Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Not planning to share IPD to other researchers

REFERENCES:
- [Background] Pal S, Myburgh J, Bansil P, Hann A, Robertson L, Gerth-Guyette E, Ambler G, Bizilj G, Kahn M, Zobrist S, Manis MR, Styke NA, Allan V, Ansbro R, Akingbade T, Bryan A, Murphy SC, Kublin JG, Layton M, Domingo GJ. Reference and point-of-care testing for G6PD deficiency: Blood disorder interference, contrived specimens, and fingerstick equivalence and precision. PLoS One. 2021 Sep 20;16(9):e0257560. doi: 10.1371/journal.pone.0257560. eCollection 2021. PMID 34543346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the Seattle Malaria Clinical Trials Center (MCTC), based at the Fred Hutch Cancer Research Center and the University of Washington.
  Participants were recruited from the greater Seattle area, and and targeted populations with expected high prevalence of glucose-6-phosphate dehydrogenase activity (G6PD) deficiency, including Southeast Asian populations and African-American populations.
Groups:
- G6PD Diagnostic Testing: Participants provided whole blood samples as well as finger-stick capillary blood samples.
  At the clinic site lab, study staff performed the Standard Diagnostics (SD) Biosensor point-of-care (POC) G6PD test assay and the POC HemoCue hemoglobin test on both finger-stick blood and whole blood samples.
  At the reference laboratory, G6PD activity was measured from whole blood samples using the Pointe Scientific G6PD reference assay and hemoglobin was measured using a hematology analyzer.
Period: Overall Study
Arm/Group | G6PD Diagnostic Testing
Started | 250
Completed | 250
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The final analytic population excludes 36 Normal G6PD Males who were selected and excluded for Threshold Determination. Additionally 1 individual was excluded because venous blood was not collected.
Groups:
- G6PD Diagnostic Testing: Participants provided whole blood samples as well as finger-stick capillary blood samples.
  At the clinic site lab, study staff performed the SD Biosensor POC G6PD test and the POC HemoCue hemoglobin test on both finger stick blood and whole blood samples.
  At the reference laboratory, G6PD activity was measured from whole blood samples using the Pointe Scientific G6PD reference assay and hemoglobin was measured using a hematology analyzer.
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (12.3)
Age, Customized [Count of Participants; unit: Participants]
  ≤ 21 years of age | 7
  22 - 64 years of age | 203
  ≥ 65 years of age | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135
  Male | 78
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 27
  Black/African American | 34
  Caucasian/White | 133
  More than one race | 15
  Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of SD Biosensor POC G6PD Test for Identifying G6PD Deficient Individuals
Description: For the purposes of this study, an individual was considered G6PD deficient if they tested positive in the Pointe Scientific assay. A true positive was defined as a participant with ≤ 30% of normal G6PD activity in circulating venous blood determined by the Pointe Scientific test.
  Diagnostic sensitivity of the SD Biosensor G6PD test is defined as the percentage of participants who tested positive for G6PD deficiency on the reference test who were identified by the test assay as positive, calculated as:
  Number of participants who were both test and true positive / (Number of participants who were test and true positive + Number of participants who were test negative but true positive [ie false negative]) * 100%.
  Sensitivity of the SD Biosensor POC G6PD test was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: The final analytic population with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 212
percentage of participants
  Venous Blood: number analyzed (Participants) | 203
  Venous Blood | 100.0 [59.0 to 100.0]
  Capillary Blood | 100.0 [59.0 to 100.0]

2. Primary Outcome: Sensitivity of SD Biosensor POC G6PD Test for Identifying Women With Intermediate G6PD Activity
Description: To investigate the performance of the SD Biosensor G6PD test to distinguish females with intermediate G6PD activity from females with normal activity, assay sensitivity was determined at a G6PD activity threshold of 70%. A true positive for intermediate G6PD activity in females was defined as G6PD activity between 30 and 70% of normal in circulating venous blood as determined by the Pointe Scientific test.
  Sensitivity of the SD Biosensor POC G6PD test is the percentage of women who tested positive for intermediate G6PD activity on the reference test who were identified by the test assay as positive, calculated as:
  Number of women who were both test and true positive / (Number of women who were test and true positive + Number of women who were test negative but true positive [ie false negative]) * 100%.
  Sensitivity of the SD Biosensor G6PD test for identifying females with intermediate G6PD activity was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: Females in the final analytic population with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- G6PD Diagnostic Testing: Participants provided whole blood samples as well as finger-stick capillary blood samples.
  At the clinic site lab, study staff performed the SD Biosensor POC G6PD test assay and the POC HemoCue hemoglobin test on both finger stick blood and whole blood samples.
  At the reference laboratory, G6PD activity was measured from whole blood samples using the Pointe Scientific G6PD reference assay and hemoglobin was measured using a hematology analyzer.
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 135
percentage of participants
  Venous Blood: number analyzed (Participants) | 133
  Venous Blood | 100.0 [39.8 to 100.0]
  Capillary Blood | 75.0 [19.4 to 99.4]

3. Primary Outcome: Specificity of SD Biosensor POC G6PD Test for Identifying G6PD Deficient Individuals
Description: For the purposes of this study, an individual was considered G6PD deficient if they tested positive by the Pointe Scientific assay. A true negative was defined as > 30% of normal G6PD activity in circulating venous blood as determined by the Pointe Scientific test.
  Specificity is the percentage of participants who tested negative for G6PD deficiency on the reference test who were identified as negative using the test assay, calculated as:
  Number of participants who were both test and true negative / (Number of participants who were test and true negative + Number of participants who were test positive but true negative [ie false positive]) * 100%.
  Specificity of the SD Biosensor G6PD test was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: The final analytic population with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 212
percentage of participants
  Venous Blood: number analyzed (Participants) | 203
  Venous Blood | 94.9 [90.8 to 97.5]
  Capillary Blood | 98.5 [95.8 to 99.7]

4. Primary Outcome: Specificity of SD Biosensor G6PD Test for Identifying Women With Intermediate G6PD Activity
Description: To investigate the performance of the SD Biosensor G6PD test to distinguish females with intermediate G6PD activity from females with normal activity, the specificity was determined at a G6PD activity threshold of 70%. A true negative for intermediate G6PD activity in females was defined as G6PD activity > 70% of normal in circulating venous blood as determined by the Pointe Scientific test.
  Specificity is the percentage of participants who tested negative for G6PD deficiency on the reference test who were identified as negative using the test assay, calculated as:
  Number of participants who were both test and true negative / (Number of participants who were test and true negative + Number of participants who were test positive but true negative [ie false positive]) * 100%.
  Specificity of the SD Biosensor G6PD test was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: Females in the final analytic population with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 135
percentage of participants
  Venous Blood: number analyzed (Participants) | 133
  Venous Blood | 83.7 [76.2 to 89.6]
  Capillary Blood | 92.4 [86.4 to 96.3]

5. Secondary Outcome: Accuracy Between the SD Biosensor POC G6PD Test Assay and the Pointe Scientific Test Kit
Description: Accuracy between the SD Biosensor POC G6PD test assay and the Pointe Scientific G6PD reference assay was calculated as the percent agreement between both G6PD tests, ie, the percentage of participants with the same diagnosis according to both tests (either deficient, intermediate, or normal G6PD levels).
  Accuracy of the SD Biosensor G6PD test was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: The final analytic population with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 212
percentage of participants
  Venous blood: number analyzed (Participants) | 203
  Venous blood | 85.7 [80.1 to 90.2]
  Capillary blood | 93.9 [89.7 to 96.7]

6. Secondary Outcome: Accuracy Between the SD Biosensor POC G6PD Test Measure of Hemoglobin and the Reference Hemoglobin Test
Description: Accuracy between the SD Biosensor POC G6PD test measure of hemoglobin and the hemoglobin reference assay was calculated as the percentage agreement between both tests, ie, the percentage of participants with the same diagnosis according to both tests (either non/mild anemia, moderate anemia or severe anemia).
Time Frame: All samples were collected on study day 1
Population: The final analytic population with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 212
percentage of participants
  Venous blood: number analyzed (Participants) | 203
  Venous blood | 97.5 [94.3 to 99.1]
  Capillary blood | 89.6 [84.7 to 93.4]

7. Secondary Outcome: Median G6PD Values Measured by the SD Biosensor G6PD Test for Venous and Capillary Blood Samples
Time Frame: All samples were collected on study day 1
Population: The final analytic population with available data
Measure: Median (Inter-Quartile Range); unit: units / gram of hemoglobin
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 213
units / gram of hemoglobin
  Venous blood: number analyzed (Participants) | 212
  Venous blood | 7.6 [6.8 to 8.5]
  Capillary blood | 6.8 [6.1 to 7.5]
Statistical Analysis 1: Comparison: G6PD Diagnostic Testing; Comparison of SD Biosensor POC G6PD test results for capillary and venous samples; Test type: Other; p < 0.001, K-sample test; The p-value was calculated using a nonparametric k-sample test on the equality of medians

ADVERSE EVENTS:
Time Frame: Approximately 30 minutes
Arm/Group | G6PD Diagnostic Testing
All-Cause Mortality (participants affected / at risk) | 0/250
Serious Adverse Events (participants affected / at risk) | 0/250
Other Adverse Events (participants affected / at risk) | 0/250

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT04010695/Prot_SAP_000.pdf